CLINICAL TRIAL: NCT04176146
Title: Accelerating the Use of Evidence-based Innovation in Health Care Systems
Brief Title: Nudging Healthcare Organizations to Adopt New Care Delivery Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amber Barnato, Professor of Health Policy and Clinical Practice and of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Dartmouth IRB protocol #28763; 1U19HS024075 (AHRQ)
Record Dates: First submitted 2019-11-14; First posted 2019-11-25 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Delivery of Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nudge Letter (Experimental): Participants receive a letter that highlights their performance vs. peer organizations on up to seven care delivery practices featured in the National Survey of Healthcare Organizations and Systems (NSHOS). The letter includes a link to access technical assistance resources and is sent alongside the participant's NSHOS respondent report.
  Interventions: Behavioral: Peer comparison and social norms messaging
- Control Letter (No Intervention): Participants receive a letter with a link to technical assistance resources; the letter is sent alongside the participant's NSHOS survey respondent report.

INTERVENTIONS:
Behavioral: Peer comparison and social norms messaging — This group will receive a letter noting that their organization has not implemented at least one common care delivery practice that a majority their peers have already implemented. The letter will also note the percentage of peer organizations that have implemented the practice. This is done using peer comparison data and social norms messaging.
  Arms: Nudge Letter

SUMMARY:
This two-arm, parallel group randomized controlled trial will assess the impact of written social norms messaging (i.e., behavioral 'nudges') on healthcare organization administrators' decision to access online resources that support the adoption of evidence-based healthcare delivery practices. The healthcare delivery practices include the use of population screening tools, clinical practice guidelines, and shared decision making training.

DETAILED DESCRIPTION:
The purpose of this study is to assess if behavioral 'nudges' impact the likelihood of healthcare organization administrators accessing technical assistance resources to support uptake of care delivery practices that: (1) have the potential to improve patient outcomes; and (2) have already been adopted by most healthcare organizations. A 'nudge' is a change in the way information is presented that attempts to steer people in a certain direction but does not restrict their choices.

The investigator will conduct a randomized controlled trial of written messages to healthcare administrators at three types of healthcare organizations - physician practices, hospitals and healthcare systems - from among 3,402 administrators who completed Dartmouth's National Survey of Healthcare Organizations and Systems (NSHOS) in 2017-2018.

In Fall 2019 the investigator will mail a customized report to all NSHOS respondents that compares their organizations' survey responses to their peer organizations. The investigator will randomize the 2,387 respondents whose organizations have not implemented one or more of up to seven chosen care delivery practices to cover letters with or without social norms messaging. The written messaging in the 'control condition' cover letter lists the practices for which the NSHOS team has prepared technical assistance materials in support of practice adoption, and contains a link to these online resources. The 'intervention condition' additionally highlights the organization's performance compared to its peers in adopting the practices using visual data display and explicit social norms messaging.

ELIGIBILITY:
Inclusion Criteria:

* Participant responded to NSHOS survey and reported that their organization had not implemented at least one of up to seven pre-determined care delivery practices, out of the following eight practices featured in the NSHOS: Screening for opioid use specifically; Screening for substance use disorders; Screening for depression; Screening for interpersonal violence; Method for identifying high-cost patients; Use of evidence-based guidelines for congestive heart failure; Use of evidence-based guidelines for sepsis (included in letters to healthcare system administrators, but not hospitals or physician practices); Training for shared decision making (included in letters to hospitals and physician practices but not healthcare systems)

Exclusion Criteria:

* Did not respond to NSHOS survey
* Participant responded to NSHOS survey and reported that their organization had already implemented each of seven pre-determined care delivery practices, out of the following eight practices featured in the NSHOS: Screening for opioid use specifically; Screening for substance use disorders; Screening for depression; Screening for interpersonal violence; Method for identifying high-cost patients; Use of evidence-based guidelines for congestive heart failure; Use of evidence-based guidelines for sepsis (included in letters to healthcare system administrators, but not hospitals or physician practices); Training for shared decision making (included in letters to hospitals and physician practices but not healthcare systems)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2387 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who access the technical assistance resource webpage | Up to 2 months after letter is sent
  The percentage of participants who access the technical assistance webpage will be determined by email and webpage analytics. The primary analysis will be intention to treat (i.e., among all participants sent a letter); a secondary analysis will be a 'per protocol' analysis (i.e., among all participants whose letter was not sent back as undeliverable). Exploratory sub-group analyses will be conducted by each strata characteristic (e.g., whether organization category influences the likelihood of accessing the webpage).

SECONDARY OUTCOMES:
Number of unique resource views on technical assistance resource webpage | Up to 2 months after letter is sent
  The number of unique resources viewed from the webpage, as determined by website analytics.
Percentage of participants who request connection to peer organizations via the technical assistance resource webpage | Up to 2 months after letter is sent
  The number of unique organizations that request to be matched with other healthcare organizations that have successfully implemented one of the care delivery practices, in order to learn from their experiences (there will be a clickable link on the webpage for organizations to request this connection). This will be determined by website analytics.
Perceived effect of letter on administrators' intentions | Up to 4 months after letter is sent
  Effect of letter on administrators' intentions and actions, measured by qualitative interviews in a sub-sample of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Amber E Barnato, MD, MPH, MS, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No